CLINICAL TRIAL: NCT03199014
Title: the Effect of Prolonged Inflation Time During Drug-eluting Stents Deployment Compared With Conventional Method for ST-elevation Myocardial Infarction
Brief Title: the Effect of Prolonged Inflation Time During Stents Deployment for ST-elevation Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WestChinaH-CVD-001
Record Dates: First submitted 2016-12-10; First posted 2017-06-26 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Acute ST-elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- prolonged deployment strategy group (Experimental): in "deploying the Drug-eluting Stents with a prolonged time" group,the inflation time was more than 30 seconds when the Drug-eluting Stents deploying,unless the patients was unstable.
  Interventions: Device: deploying the Drug-eluting Stents with a prolonged time
- rapid deployment strategy group (Active Comparator): in "deploying the Drug-eluting Stents with a conventional time" group, a conventional method was used to deploying drug-eluting stents,the actual inflation time was within 10s determined by interventional cardiologist.
  Interventions: Device: deploying the Drug-eluting Stents with a conventional time

INTERVENTIONS:
Device: deploying the Drug-eluting Stents with a prolonged time — the inflation time was more than 30 seconds when the Drug-eluting Stents deploying.The PROMUS Element Plus Stent or Co-Cr sirolimus-eluting coronary stent system（GuReater）was used in this study
  Arms: prolonged deployment strategy group
Device: deploying the Drug-eluting Stents with a conventional time — the actual inflation time was within 10s determined by interventional cardiologist.The PROMUS Element Plus Stent or Co-Cr sirolimus-eluting coronary stent system（GuReater）was used in this study
  Arms: rapid deployment strategy group

SUMMARY:
The purpose of this study is to determine whether prolonged inflation time on drug-eluting stents deployment for ST-elevation myocardial Infarction was better than conventional stents deployment.

ELIGIBILITY:
Inclusion Criteria:

* men and women ≥18 years with ST-elevation Myocardial Infarction;
* patients with STEMI and ischemic symptoms of less than 12 hours'duration;
* patients with STEMI and ischemic symptoms of less than 12 hours' duration who have contraindications to fibrinolytic therapy, irrespective of the time delay from FMC;
* patients with STEMI if there is clinical and/or ECG evidence of ongoing ischemia between 12 and 24 hours after symptom onset;
* when angiography was completed, guide wire could cross the lesion in the culprit vessel, TIMI≥1，with feasibility to direct stenting

Exclusion Criteria:

* cardiac shock, or acute severe heart failure;
* the lesion was highly calcified, excessive proximal tortuosity,left main artery lesion, restenosis lesion,vein graft lesion,total occlusions;
* True bifurcation lesions;
* Stenosis≤50% and TIMI flow grade 3;
* history of PCI in target vessel;
* diameter of the target vessel less than 2 mm;
* severe liver and kidney dysfunction;
* inability to give informed written consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With TIMI 3 | 1 minute after sent was deployed
  TIMI 0 flow (no perfusion) refers to the absence of any antegrade flow beyond a coronary occlusion.TIMI 1 flow (penetration without perfusion) is faint antegrade coronary flow beyond the occlusion, with incomplete filling of the distal coronary bed.TIMI 2 flow (partial reperfusion) is delayed or sluggish antegrade flow with complete filling of the distal territory.TIMI 3 is normal flow which fills the distal coronary bed completely
corrected TIMI frame count(frames) | 1 minute after sent was deployed
  Grading was done on cinefilm at 15frames/s made in a Philips digital coronary imaging catheterization laboratory.
myocardial blush grade | 1 minute after sent was deployed
  0, no myocardial blush or contrast density; 1, minimal myocardial blush or contrast density; 2,moderate myocardial blush or contrast density but less than that obtained during angiography of a contralateral or ipsilateral non- infarct-related coronary artery; and 3, normal myocardial blush or contrast density, comparable with that obtained during angiography of a contralateral or ipsilateral non-infarct-related coronary artery

SECONDARY OUTCOMES:
Number of Participants ST-segment resolution | 60min after the operation
  1, normalized, defined as no residual ST-segment elevation; 2, improved, defined as a residual ST-segment elevation ,70% of with that on the first ECG; and 3, unchanged, defined as a residual ST-segment elevation 70% of that on the first ECG
Number of Participants Death from cardiac causes | one month after the operation
  death from acute myocardial infarction, cardiac perforation, or pericardial tamponade; an arrhythmia or conduction abnormality; complications of the interventional procedure at baseline
Number of Participants Target-vessel revascularization | one month after the operation
  any revascularization intervention (PCI or CABG) occurring in a treated vessel at any time after the index intervention.
Number of Participants stent thrombosis | one month after the operation
  evidence of any myocardial infarction with angiographic confirmation of in-stent thrombus or unexplained death within 30 days after the procedure as stent thrombosis
Number of Participants had Major bleeding | one month after the operation
  any symptomatic intracranial hemorrhage, or clinically overt signs of hemorrhage (including imaging) associated with a drop in hemoglobin of>= g/dL (or when the hemoglobin concentration is not available, an absolute drop in hematocrit of>=15%)

OTHER OUTCOMES:
Procedural time | form start puncturing vascular until the operation was completed intraoperative
  minute
Radiation exposure time | form start puncturing vascular until the operation was completed intraoperative
  minute

CONTACTS AND LOCATIONS:
Overall Officials: He yong, Study Director — west china hospital of sichuan univercity
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sabatier R, Hamon M, Zhao QM, Burzotta F, Lecluse E, Valette B, Grollier G. Could direct stenting reduce no-reflow in acute coronary syndromes? A randomized pilot study. Am Heart J. 2002 Jun;143(6):1027-32. doi: 10.1067/mhj.2002.122509. PMID 12075259
- [Background] Ozdemir R, Sezgin AT, Barutcu I, Topal E, Gullu H, Acikgoz N. Comparison of direct stenting versus conventional stent implantation on blood flow in patients with ST-segment elevation myocardial infarction. Angiology. 2006 Aug-Sep;57(4):453-8. doi: 10.1177/0003319706290620. PMID 17022381
- [Background] Li C, Zhang B, Li M, Liu J, Wang L, Liu Y, Wang Z, Wen S. Comparing Direct Stenting With Conventional Stenting in Patients With Acute Coronary Syndromes: A Meta-Analysis of 12 Clinical Trials. Angiology. 2016 Apr;67(4):317-25. doi: 10.1177/0003319715585662. Epub 2015 May 11. PMID 25964649
- [Background] Hovasse T, Mylotte D, Garot P, Salvatella N, Morice MC, Chevalier B, Pichard A, Lefevre T. Duration of balloon inflation for optimal stent deployment: five seconds is not enough. Catheter Cardiovasc Interv. 2013 Feb;81(3):446-53. doi: 10.1002/ccd.23343. Epub 2012 Jan 10. PMID 22109977
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Gibson CM, Murphy SA, Rizzo MJ, Ryan KA, Marble SJ, McCabe CH, Cannon CP, Van de Werf F, Braunwald E. Relationship between TIMI frame count and clinical outcomes after thrombolytic administration. Thrombolysis In Myocardial Infarction (TIMI) Study Group. Circulation. 1999 Apr 20;99(15):1945-50. doi: 10.1161/01.cir.99.15.1945. PMID 10208996
- [Background] Gibson CM, Cannon CP, Daley WL, Dodge JT Jr, Alexander B Jr, Marble SJ, McCabe CH, Raymond L, Fortin T, Poole WK, Braunwald E. TIMI frame count: a quantitative method of assessing coronary artery flow. Circulation. 1996 Mar 1;93(5):879-88. doi: 10.1161/01.cir.93.5.879. PMID 8598078
- [Derived] Ma M, Wang L, Diao KY, Liang SC, Zhu Y, Wang H, Wang M, Zhang L, Yang ZG, He Y. A randomized controlled clinical trial of prolonged balloon inflation during stent deployment strategy in primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: a pilot study. BMC Cardiovasc Disord. 2022 Feb 4;22(1):30. doi: 10.1186/s12872-022-02477-0. PMID 35120436